CLINICAL TRIAL: NCT02821416
Title: A Double-Blind, Randomized, Parallel Group, Placebo-Controlled Multi-Centre Study to Evaluate the Effect of Benralizumab on Allergen-Induced Inflammation in Mild, Atopic Asthmatics
Brief Title: Study to Evaluate the Effect of Benralizumab on Allergen-Induced Inflammation in Mild, Atopic Asthmatics
Acronym: ARIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3250C00040
Record Dates: First submitted 2016-06-17; First posted 2016-07-01 (Estimated); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benralizumab (Experimental): Benralizumab administered subcutaneously
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab subcutaneously on study day 0 until study week 16 day 1 inclusive
  Arms: Benralizumab
Other: Placebo — Placebo subcutaneously on study week 0 until study week 16 day 1 inclusive
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, parallel group, placebo-controlled study designed to evaluate the effect of a fixed 30 mg dose of benralizumab administered subcutaneously every 4 weeks on allergen-induced inflammation in subjects with mild atopic asthma challenged with an inhaled allergen.

DETAILED DESCRIPTION:
This randomized, double-blind, parallel group, placebo-controlled study will evaluate the effect of a fixed 30 mg dose of benralizumab administered subcutaneously every 4 weeks for 3 doses on allergen-induced inflammation in subjects with mild atopic asthma challenged with an inhaled allergen.

Approximately 38 non-smoking men and women (18 - 65 years of age) corticosteroid-free (oral and inhaled) mild, atopic asthmatics who have demonstrated a dual (early and late) asthmatic response to inhaled allergen challenge at screening will be recruited to complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female or male aged 18 to 65 years, inclusively, at the time of enrolment.
3. General good health
4. Mild, stable, allergic asthma and asthma therapy limited to inhaled, short-acting beta 2 agonists (not more than twice weekly)
5. Positive skin-prick test to at least one common aeroallergen

Exclusion Criteria:

1. Current lung disease other than mild allergic asthma
2. Any history or symptoms of disease, including, but not limited to, cardiovascular, neurologic, autoimmune or haematologic
3. Any clinically significant abnormal findings in laboratory test results in complete blood count, coagulation, chemistry panel and urinalysis at enrolment and during screening period
4. History of anaphylaxis to any biologic therapy or vaccine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan

REFERENCES:
- See also: The CSP redacted. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00040&attachmentIdentifier=38fb2b0f-090e-4f1a-bfa3-f74c5941c69e&fileName=d3250c00040-csp-4_-_Redacted_(1).pdf&versionIdentifier=
- See also: The SAP redacted. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00040&attachmentIdentifier=d3ca7f3e-fb89-4822-97f4-85610a3f79cd&fileName=d3250c00040-sap-v2_-_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Benra 30mg q.4 Week: Benralizumab 30mg every 4 Weeks
- Placebo: Placebo every 4 Weeks
Period: Overall Study
Arm/Group | Benra 30mg q.4 Week | Placebo
Started | 23 | 23
Completed | 20 | 22
Not Completed | 3 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benra 30mg q.4 Week | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.4 (12.3) | 31.5 (13.3) | 30.9 (12.7)
Age, Customized [Count of Participants; unit: Participants]
  >=18 - <=50 | 20 | 20 | 40
  >50 - <=65 | 3 | 3 | 6
  >65 - <=75 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 9 | 3 | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 16 | 19 | 35
  Black or African American | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent of Eosinophils in Sputum 7 Hours Post Allergen Challenge
Description: To evaluate the effect of benralizumab on allergen-induced increases in eosinophils in induced sputum
Time Frame: From prechallenge to 7 hours post allergen challenge during week 9
Population: Primary Efficacy Analysis
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- Benra 30mg q.4 Weeks: Benralizumab 30 mg every 4 Weeks
Arm/Group | Benra 30mg q.4 Weeks | Placebo
Number analyzed (Participants) | 23 | 22
Percent | 0.822 (4.054) | 6.468 (9.560)
Statistical Analysis 1: Comparison: Benra 30mg q.4 Weeks vs Placebo; Test type: Superiority; p = 0.0208, Mixed Models Analysis; Model includes covariates of treatment, time post-allergen challenge , treatment*time post-allergen challenge, allergen induced at screening; Median Difference (Final Values) = -5.81, 95% CI 2-sided [-10.69 to -0.94]

2. Primary Outcome: Maximal Percentage Decrease in Forced Expiratory Volume in 1 Second 3-7 Hours Post Allergen Challenge
Description: To evaluate the effect of benralizumab on the allergen-induced late (3-7 hours post challenge) asthmatic response (LAR)
Time Frame: From prechallenge to 3 to 7 hours post allergen challenge during week 9
Population: Primary Efficacy Analysis
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- Benra 30mg q.4 Weeks: Benralizumab 30mg every 4 weeks
Arm/Group | Benra 30mg q.4 Weeks | Placebo
Number analyzed (Participants) | 23 | 22
Percent | 15.152 (8.834) | 16.275 (10.235)
Statistical Analysis 1: Comparison: Benra 30mg q.4 Weeks vs Placebo; Test type: Superiority; p = 0.3630, Mixed Models Analysis; Model includes covariates of treatment, maximum percent decrease in FEV1 late asthma response; Median Difference (Final Values) = 2.535, 95% CI 2-sided [-3.045 to 8.116]

ADVERSE EVENTS:
Time Frame: From Visit 1a to Visit 17
Arm/Group | Benra 30mg q.4 Week | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 7/23 | 14/23
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30mg q.4 Week (N=23) | Placebo (N=23)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (3)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Migraine (Nervous system disorders) | 1 (2) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (3)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This allergen challenge study was conducted in a mild, atopic asthma patient population, distinct from the current approved severe eosinophilic asthma indication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT02821416/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT02821416/SAP_001.pdf